CLINICAL TRIAL: NCT04436822
Title: Evaluation of Updated Continuous Glucose Monitoring (CGM) Form Factor in Adults, Adolescents and Pediatrics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Diabetes (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CIP330
Record Dates: First submitted 2020-06-12; First posted 2020-06-18 (Actual); Results first posted 2023-06-02 (Actual); Last update posted 2023-06-02 (Actual); Status verified 2023-05

CONDITIONS: Type 1 Diabetes Mellitus; Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2 | interventions — Continuous Glucose Monitoring

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Subjects with diabetes wearing DS5 (Experimental): Subjects wearing DS5 over 7 days and participating in FSTs.
  Interventions: Device: Continuous Glucose Monitoring

INTERVENTIONS:
Device: Continuous Glucose Monitoring — CGM and frequent sample testing

SUMMARY:
The purpose of this study is to demonstrate the performance of the Disposable Sensor (DS5) in subjects age 2 - 80 years, for the span of 170 hours (7 days).

DETAILED DESCRIPTION:
The purpose of this study is to demonstrate the performance of the Disposable Sensor (DS5) in subjects age 2 - 80 years, for the span of 170 hours (7 days).

This is a multi-center study.

ELIGIBILITY:
Inclusion Criteria:

1. Individual is 2 - 80 years of age at time of enrollment.
2. Subject has a clinical diagnosis of type 1 or type 2 diabetes:

   1. If subject is 14-80 years of age, subject has a clinical diagnosis of type 1 or type 2 diabetes for a minimum of 6 months duration as determined via medical record/ source documentation by an individual qualified to make a medical diagnosis.
   2. If subject is 2-13 years of age, subject has a clinical diagnosis of type 1 or type 2 diabetes as determined via medical record/ source documentation by an individual qualified to make a medical diagnosis.
3. If subject is participating in YSI™* FST , subject has adequate venous access as assessed by investigator or appropriate staff.
4. Subjects participating in the high and low glucose challenges must have an insulin carbohydrate ratio(s) and insulin sensitivity factor(s). Subjects without ratios may participate under observation only.

Exclusion Criteria:

1. Subject will not tolerate tape adhesive in the area of sensor placement as assessed by a qualified individual.
2. Subject has any unresolved adverse skin condition in the area of sensor or device placement (e.g., psoriasis, rash, Staphylococcus infection).
3. Subject is actively participating in an investigational study (e.g., drug or device) wherein he/she has received treatment from an investigational study (drug or device) in the last 2 weeks prior to Visit 1. (Please note participation in an observational study is acceptable.)
4. Subject is female of child-bearing potential and has a pregnancy screening test that is positive.
5. Subject is a sexually active female of child-bearing potential and is not using a form of contraception deemed reliable by investigator.
6. Subject is female and plans to become pregnant during the course of the study.
7. Subject has had a hypoglycemic seizure within the past 6 months prior to enrollment.
8. Subject has had hypoglycemia resulting in loss of consciousness within the past 6 months prior to enrollment.
9. Subject has had an episode of diabetic ketoacidosis (DKA) within the past 6 months prior to enrollment.
10. Subject has a history of a seizure disorder.
11. Subject has central nervous system or cardiac disorder resulting in syncope.
12. Subject has a history of myocardial infarction, unstable angina, coronary artery bypass surgery, coronary artery stenting, transient ischemic attack (TIA), cerebrovascular accident (CVA), angina, congestive heart failure, ventricular rhythm disturbances or thromboembolic disease
13. If subject is 7-80 years of age, subject has a hematocrit (Hct) more than 10% below the lower limit of normal reference range (please note that patients may use prior blood draw from routine care as long as done within 6 months of screening and report of lab placed with subject source documents).
14. Subject has a history of adrenal insufficiency.
15. Subject is a member of the research staff involved with the study.

Ages: 2 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 317 (Actual)
Dates: Start 2020-07-15 (Actual); Primary Completion 2022-04-12 (Actual); Study Completion 2022-04-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (18):
- United States (13):
  - AMCR Institute, Escondido, California
  - Sansum Diabetes Research Institute, Santa Barbara, California
  - SoCal Diabetes, Torrance, California
  - Diablo Clinical Research, Inc., Walnut Creek, California
  - Barbara Davis Center for Childhood Diabetes, Aurora, Colorado
  - Barbara Davis Center for Diabetes, Aurora, Colorado
  - University of South Florida, Tampa, Florida
  - Atlanta Diabetes Associates, Atlanta, Georgia
  - Rocky Mountain Diabetes and Osteoporosis Center, Idaho Falls, Idaho
  - AM Diabetes and Endocrinology Center, Bartlett, Tennessee
  - Texas Diabetes & Endocrinology, Austin, Texas
  - University of Virginia Center for Diabetes Technology, Charlottesville, Virginia
  - Rainier Clinical Research Center, Inc., Renton, Washington
- China (5):
  - Nanjing First Hospital, Nanjing, Jiangsu
  - Dalian Municiple Central Hospital, Dalian, Liaoning
  - Shanghai Sixth People's Hospital, Shanghai, Shanghai Municipality
  - Children's Hospital of Fudan University, Shanghai, Shanghai Municipality
  - The Children's Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 317 subjects (175 adult subjects, 141 pediatric subjects, and 1 age-unknown subject) consented and enrolled in the overall study. Of them, 7 subjects were screening failure and 310 subjects (172 adult subjects and 138 pediatric subjects) participated in the study.
Groups:
- Adult Subjects (Age 18-80) Wearing DS5: Adult subjects (age 18-80) wearing DS5 over 7 days: Continuous Glucose Monitoring and frequent sample testing
- Pediatric Subjects (Age 2-17) Wearing DS5: Pediatric subjects (age 2-17) wearing DS5 over 7 days: Continuous Glucose Monitoring and frequent sample testing
Period: Overall Study
Arm/Group | Adult Subjects (Age 18-80) Wearing DS5 | Pediatric Subjects (Age 2-17) Wearing DS5
Started | 172 | 138
Completed | 160 | 132
Not Completed | 12 | 6
Not completed — Physician Decision | 2 | 0
Not completed — Sponsor request | 1 | 0
Not completed — Withdrawal by parent/guardian | 0 | 3
Not completed — Unsuccessful procedure | 0 | 1
Not completed — Withdrawal due to Covid-19 | 8 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — The sponsor was not able to provide the investigational product | 0 | 1

BASELINE CHARACTERISTICS:
Population: Demographics and other baseline characteristics were documented for eligible subjects (i.e., subjects who passed screening).
Groups:
- Total: Total of all reporting groups
Arm/Group | Adult Subjects (Age 18-80) Wearing DS5 | Pediatric Subjects (Age 2-17) Wearing DS5 | Total
Number analyzed (Participants) | 172 | 138 | 310
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.3 (16.8) | 10.5 (4.8) | 30.3 (22.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 78 | 60 | 138
  Male | 94 | 78 | 172
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 20 | 10 | 30
  Not Hispanic or Latino | 98 | 106 | 204
  Unknown or Not Reported | 54 | 22 | 76
Region of Enrollment [Number; unit: participants]
  United States | 121 | 117 | 238
  China | 51 | 21 | 72
BMI (kg/m2) [Mean (Standard Deviation); unit: kg/m^2] | 28.7 (6.4) | 19.8 (4.2) | 24.8 (7.1)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Readings Within 20% Agreement
Description: Mean of daily percentage of sensor values within 20% of Yellow Springs Instrument (YSI™*) reference value (within 20 mg/dL [1.1 mmol/L] when sensor values < 80 mg/dL) [4.4 mmol/L]) by age groups and DS5 insertion locations. Note Self-Monitoring Blood Glucose (SMBG) was used for age 2-6, instead of YSI. Zero calibration sensor algorithm applied to raw sensor data.
Time Frame: 7 days (170 hours)
Population: Subjects with at least 1 sensor-YSI (or sensor-SMBG for subjects 2-6 years) paired point during the sensor wear
Measure: Mean (90% Confidence Interval); unit: percentage of readings
Groups:
- Adult Subjects (Age 18-80) Wearing DS5 on the Arm: Adult subjects (age 18-80) wearing DS5 on the arm over 7 days: Continuous Glucose Monitoring and frequent sample testing. Zero calibration sensor algorithm applied to raw sensor data.
- Pediatric Subjects (Age 2-17) Wearing DS5 on the Arm: Pediatric subjects (age 2-17) wearing DS5 on the arm over 7 days: Continuous Glucose Monitoring and frequent sample testing. Zero calibration sensor algorithm applied to raw sensor data.
- Pediatric Subjects (Age 2-17) Wearing DS5 on the Buttock: Pediatric subjects (age 2-17) wearing DS5 on the buttock over 7 days: Continuous Glucose Monitoring and frequent sample testing. Zero calibration sensor algorithm applied to raw sensor data.
Arm/Group | Adult Subjects (Age 18-80) Wearing DS5 on the Arm | Pediatric Subjects (Age 2-17) Wearing DS5 on the Arm | Pediatric Subjects (Age 2-17) Wearing DS5 on the Buttock
Number analyzed (Participants) | 155 | 127 | 118
percentage of readings | 88.9 [87.1 to 90.7] | 87.5 [85.4 to 89.7] | 87.9 [85.8 to 89.9]
Statistical Analysis 1: Comparison: Adult Subjects (Age 18-80) Wearing DS5 on the Arm; Test type: Superiority; p < 0.05, ANCOVA; A generalized estimating equation model was used, considering correlation structure of day of sensor wear (1-7); Intercept from ANCOVA as agreement rate = 88.9, 90% CI 2-sided [87.1 to 90.7]
Statistical Analysis 2: Comparison: Pediatric Subjects (Age 2-17) Wearing DS5 on the Arm; Test type: Superiority; p < 0.05, ANCOVA; A generalized estimating equation model was used, considering correlation structure of day of sensor wear (1-7); Intercept from ANCOVA as agreement rate = 87.5, 90% CI 2-sided [85.4 to 89.7]
Statistical Analysis 3: Comparison: Pediatric Subjects (Age 2-17) Wearing DS5 on the Buttock; Test type: Superiority; p < 0.05, ANCOVA; A generalized estimating equation model was used, considering correlation structure of day of sensor wear (1-7); Intercept from ANCOVA as agreement rate = 87.9, 90% CI 2-sided [85.8 to 89.9]

ADVERSE EVENTS:
Time Frame: Throughout the course of the study, up to approximately 90 days (including an up to 7-day training period and a 7-day study period)
Arm/Group | Adult Subjects (Age 18-80) Wearing DS5 | Pediatric Subjects (Age 2-17) Wearing DS5
All-Cause Mortality (participants affected / at risk) | 0/172 | 0/138
Serious Adverse Events (participants affected / at risk) | 1/172 | 0/138
Other Adverse Events (participants affected / at risk) | 27/172 | 23/138
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adult Subjects (Age 18-80) Wearing DS5 (N=172) | Pediatric Subjects (Age 2-17) Wearing DS5 (N=138)
BILATERAL HYDRONEPHROSIS (Renal and urinary disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adult Subjects (Age 18-80) Wearing DS5 (N=172) | Pediatric Subjects (Age 2-17) Wearing DS5 (N=138)
Alcoholic ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arteriosclerosis (Vascular disorders) | 2 (2) | 0 (0)
Asymptomatic bacteriuria (Infections and infestations) | 1 (1) | 0 (0)
Autoimmune thyroiditis (Endocrine disorders) | 2 (2) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 5 (5) | 0 (0)
Blood potassium decreased (Investigations) | 1 (1) | 0 (0)
Carotid arteriosclerosis (Nervous system disorders) | 7 (7) | 0 (0)
Cerebral artery occlusion (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral artery stenosis (Nervous system disorders) | 1 (1) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 1 (1)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Diabetic ketosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Diabetic nephropathy (Renal and urinary disorders) | 2 (2) | 0 (0)
Diabetic neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Dry eye (Eye disorders) | 1 (1) | 0 (0)
Dyslipidaemia (Metabolism and nutrition disorders) | 6 (6) | 0 (0)
Gallbladder polyp (Hepatobiliary disorders) | 3 (3) | 0 (0)
Giant cell tumour of tendon sheath (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Growth retardation (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Helicobacter gastritis (Infections and infestations) | 0 (0) | 1 (1)
Hepatic cyst (Hepatobiliary disorders) | 3 (3) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic mass (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic steatosis (Hepatobiliary disorders) | 5 (5) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Infusion site infection (Infections and infestations) | 0 (0) | 1 (1)
Infusion site pain (General disorders) | 0 (0) | 2 (2)
Ketosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Left atrial enlargement (Cardiac disorders) | 1 (1) | 0 (0)
Medical device site bruise (General disorders) | 0 (0) | 1 (1)
Medical device site pain (General disorders) | 0 (0) | 1 (4)
Medical device site rash (General disorders) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 3 (3) | 0 (0)
Non-alcoholic fatty liver (Hepatobiliary disorders) | 1 (1) | 0 (0)
Otitis media (Infections and infestations) | 0 (0) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 4 (4) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Pleural mesothelioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Poor quality sleep (Psychiatric disorders) | 1 (1) | 0 (0)
Postoperative wound infection (Infections and infestations) | 1 (1) | 0 (0)
Prostatic calcification (Reproductive system and breast disorders) | 3 (3) | 0 (0)
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Renal cyst (Renal and urinary disorders) | 5 (5) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1)
Serum ferritin decreased (Investigations) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 1 (1) | 0 (0)
Thyroid mass (Endocrine disorders) | 5 (5) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 5 (5)
Urinary tract infection (Infections and infestations) | 2 (2) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Vitamin D decreased (Investigations) | 2 (2) | 0 (0)
Vitamin D deficiency (Metabolism and nutrition disorders) | 4 (4) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (2) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2022-03-31): https://cdn.clinicaltrials.gov/large-docs/22/NCT04436822/Prot_000.pdf
  • Statistical Analysis Plan (2022-03-31): https://cdn.clinicaltrials.gov/large-docs/22/NCT04436822/SAP_001.pdf